CLINICAL TRIAL: NCT05201690
Title: A Randomized, Double-blinded, Placebo-controlled, Phase I Clinical Trial to Evaluate the Safety, Tolerability and Pharmacokinetic Profiles of VV116 After Multiple Ascending Doses Administered Orally to Chinese Healthy Volunteers
Brief Title: Safety and Pharmacokinetics Study of Multiple Ascending Doses of VV116 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: VV116-02
Record Dates: First submitted 2021-12-29; First posted 2022-01-21 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2021-12

CONDITIONS: Healthy Subjects
Keywords: VV116; Phase I; dose-escalation; Healthy Volunteers; Safety; Tolerability; Pharmacokinetic
MeSH Terms: interventions — GS-621763; Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VV116 200 mg Group (Experimental): VV116 200 mg Group
  Interventions: Drug: VV116 200 mg Group
- VV116 400 mg Group (Experimental): VV116 400 mg Group
  Interventions: Drug: VV116 400mg Group
- VV116 600 mg Group (Experimental): VV116 600 mg Group
  Interventions: Drug: VV116 600mg Group
- Placebo (Placebo Comparator): VV116 Matching placebo tablets; Multiple doses
  Interventions: Drug: VV116 200 mg Group; Drug: VV116 400mg Group; Drug: VV116 600mg Group

INTERVENTIONS:
Drug: VV116 200 mg Group — Drug: VV116 9 subjects will receive VV116 200 mg, orally, QD12h, 5.5 days ;
  Arms: Placebo; VV116 200 mg Group
Drug: VV116 400mg Group — Drug: VV116 9 subjects will receive VV116 400 mg, orally, QD12h, 5.5 days ;
  Arms: Placebo; VV116 400 mg Group
Drug: VV116 600mg Group — Drug: VV116 9 subjects will receive VV116 600 mg, orally, QD12h, 5.5 days ;
  Arms: Placebo; VV116 600 mg Group

SUMMARY:
This is a randomized, double-blinded, placebo-controlled, single-center phase I clinical trial. The objective of this study is to evaluate the safety, tolerability, pharmacokinetic profiles of VV116 tablets after multiple ascending doses administered orally to Chinese healthy volunteers.

DETAILED DESCRIPTION:
Multiple-dose ascending design is used in the trial, VV116/Placebo is administered sequentially from low-dose to high-dose and each subject can only orally receive one dose level. There are 3 dose groups (200mg, 400mg, 600mg), investigational product is orally administrated BID for 5.5 days, the last dose is taken in D6 morning. When 7th day visit after last dose (D12) is completed for previous dose group, investigator and sponsor will evaluate the safety and determine whether the next dose group can be started. 12 subjects will be enrolled in each dose group and the ratio of investigational product to placebo is 3:1.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects between the ages of 18 and 45 years;
2. Body weight no less than 50 kg for male, no less than 45 kg for female; Body Mass Index of 19 to 26kg/m2;
3. Physical examination, vital signs examination, laboratory examination, ECG, B-ultrasound and fundus examination results were normal or abnormal without clinical significant;
4. Subjects who are willing to take proper contraceptive during the study and within 3 months after the study completed;
5. Subjects who are able to understand and follow study plans and instructions; Subjects who have voluntarily decided to participate in this study, and signed the informed consent form;

Exclusion Criteria:

1. Subjects with hypersensitivity to VV116 or any of the excipients;
2. Subjects with allergic diseases or allergic constitution;
3. Subjects with central nervous system,cardiovascular system,gastrointestinal, respiratory system,urinary,Hematologic System,metabolic disorders that require medical intervention or other diseases (such as psychiatric history) that are not suitable for clinical trials;
4. Blood donation or blood loss ≥ 400 mL within 3 months prior to inclusion, or have a history of blood product use history;
5. Participated in a clinical study involving another investigational drug within 3 month before the screening visit;
6. Taken any prescription drugs, non-prescription drugs, Chinese herbal medicine or health care products within 2 weeks prior to screening;
7. Drug or alcohol addicts within 1 year prior to screening, who drink at least twice a day or more than 14 units per week, or who are addicted to alcohol (1 unit ≈200 mL beer with 5% alcohol content, 25 mL spirits with 40% alcohol content or 85 mL wine with 12% alcohol content) ;
8. Those who smoke more than 10 cigarettes per day and do not agree to avoid using any tobacco products during the trial period;
9. Those who cannot quit smoking or drinking during the trial;
10. Those who are positive for hepatitis B surface antigen (HBsAg), HCV antibody, syphilis antibody and HIV antibody;
11. Abnormal and clinically significant chest radiographs (anteroposterior);
12. B ultrasound examination showed moderate to severe fatty liver;
13. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) exceeded the upper normal limit (ULN) at screening time or baseline;
14. Glomerular filtration rate (eGFR) < 90 mL/min/1.73m2 at screening time or baseline;
15. Abnormal ecg at screening or baseline, single QTcF (corrected for heart rate) > 450 ms in men, > 470 ms in women, and/or other clinically significant abnormalities;
16. Pregnant or lactating women or male subjects whose spouse has a child care plan within 3 months;
17. The investigator believes that there are other factors that are not suitable for participating in this trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-01-23 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment emergent treatment-related adverse event(s) | Dosing through follow-up call (7 days after last dose of investigational product)
  Frequency, severity and causal relationship of treatment emergent adverse events (TEAEs) and withdrawals due to TEAEs
Number of participants with laboratory test findings of potential clinical importance | Dosing through follow-up call (7 days after last dose of investigational product)
Number of participants with vital signs findings of potential clinical importance | Dosing through follow-up call (7 days after last dose of investigational product)
Number of participants with ECG findings of potential clinical importance | Dosing through follow-up call (7 days after last dose of investigational product)
  Number of subjects with change from baseline in electrocardiogram (ECG) parameters

SECONDARY OUTCOMES:
Tmax | Calculated using concentration data collected from predose to 48 hours postdose
  Time to reach maximum observed plasma concentration
Cmax | Calculated using concentration data collected from predose to 48 hours postdose
  Maximum observed plasma concentration
T1/2 | Calculated using concentration data collected from predose to 48 hours postdose
  Terminal half life
AUC0-T | Area under the serum concentration time profile from time zero to the time of the last quantifiable concentration.
  Calculated using concentration data collected from predose to 48 hours postdose
AUC0-∞ | Calculated using concentration data collected from predose to 48 hours postdose
  Area under the plasma concentration-time curve from time 0 extrapolated to infinity

CONTACTS AND LOCATIONS:
Overall Officials: Gangyi Liu, Principal Investigator — Shanghai Xuhui Central Hospital
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, China